CLINICAL TRIAL: NCT02128230
Title: A Phase II Trial For High-Risk Myeloma Evaluating Accelerating and Sustaining Complete Remission (AS-CR) by Applying Non-Host-Exhausting and Timely Dose-Reduced Mel-80-CFZ-TD-Pace Transplant(s) With Interspersed Mel-20-CFZ-TD-Pace With CFZ-RD and CFZ-D Maintenance
Brief Title: UARK 2012-02 Trial For High-Risk Myeloma Evaluating Accelerating and Sustaining Complete Remission
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment and Futility as determined by Amgen's Carfilzomib NASCR program.
Sponsor: University of Arkansas (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 134668
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma
Keywords: High-Risk; Carfilzomib
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; carfilzomib; Thalidomide; Dexamethasone; Calcium Dobesilate; Cisplatin; Doxorubicin; Cyclophosphamide; Etoposide; Granulocyte Colony-Stimulating Factor; Filgrastim; Biological Products; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Total Therapy 5b (Experimental): Induction, optional bridging, first transplant, optional bridging, inter-therapy, optional bridging, second transplant, optional bridging, consolidation, maintenance
  Interventions: Device: myPRS; Drug: Induction 1 - MEL-10+CFZ-TD-PACE; Drug: First Transplant - MEL-80+CFZ-TD-PACE + PBSC (biologic); Drug: Inter-Therapy - MEL-20+CFZ-TD-PACE (75%); Drug: Second Transplant - MEL-80+CFZ-TD-PACE + PBSC (biologic); Drug: Consolidation - CFZ-TD-PACE; Drug: Maintenance - CFZ-R(T)-D

INTERVENTIONS:
Device: myPRS — Genome expression profiling used to identify high-risk and low-risk multiple myeloma
  Other Names: Gep70
Drug: Induction 1 - MEL-10+CFZ-TD-PACE — Melphalan (MEL) and Carfilzomib (CFZ) will be given into a central venous catheter. Thalidomide (T) is a capsule and Dexamethasone (D) is a pill; both will be taken by mouth. Cisplatin (P), Adriamycin (A), Cyclophosphamide (C) and Etoposide (E) are all given into the vein (IV) by a continuous infusion through a central catheter. After completion of the continuous chemotherapy, Granulocyte colony-stimulating factor (G-CSF), a shot just under the skin to help the bone marrow and blood counts recover more quickly after chemotherapy, will be given.
  Regimen: CFZ 20 mg/m2 on days 1, 5, & 6; MEL 10mg/m2 on day 3; T 200 mg/d, D 40 mg/d, P 10 mg/m2/d, A 10 mg/m2/d, C 400 mg/m2/d, and E 40 mg/m2/d on days 5-8; G-CSF 10 mcg/kg/day from day 11 through end of Peripheral Blood Stem Cell (PBSC) collection.
  Optional Bridging with T 50 mg/d and D 20 mg on day 1-4 every 21 days until 1st transplant.
  Other Names: Melphalan (Alkeran™); Carfilzomib (Kyprolis®); Thalidomide (Thalomid®); Dexamethasone (Decadron®); Cisplatin (CDDP) (Platinol®); Doxorubicin (Adriamycin®); Cyclophosphamide (Cytoxan®); Etoposide (VP-16) (Vepesid®); Granulocyte colony-stimulating factor (G-CSF), filgrastim (Neupogen®)
Drug: First Transplant - MEL-80+CFZ-TD-PACE + PBSC (biologic) — Melphalan (MEL) and Carfilzomib (CFZ) will be given into a central venous catheter. Thalidomide (T) is a capsule and Dexamethasone (D) is a pill; both will be taken by mouth. Cisplatin (P), Adriamycin (A), Cyclophosphamide (C) and Etoposide (E) are all given into the vein (IV) by a continuous infusion through a central catheter. After completion of the continuous chemotherapy, Granulocyte colony-stimulating factor (G-CSF), a shot just under the skin to help the bone marrow and blood counts recover more quickly after chemotherapy, will be given.
  Regimen: CFZ 20 mg/m2 on days -5 & -4; MEL 20 mg/m2/d, T 200 mg/d, D 40 mg/d, P 10 mg/m2/d, A 10 mg/m2/d, C 100 mg/m2/d, and E 80 mg/m2/d on days -5 & -2; PBSC transplant on day 0.
  Optional Bridging with T 50 mg/d and D 20 mg on day 1-4 every 21 days until inter-therapy.
  Other Names: Autologous Peripheral Blood Stem Cell Transplant; Melphalan (Alkeran™); Carfilzomib (Kyprolis®); Thalidomide (Thalomid®); Dexamethasone (Decadron®); Cisplatin (CDDP) (Platinol®); Doxorubicin (Adriamycin®); Cyclophosphamide (Cytoxan®); Etoposide (VP-16) (Vepesid®)
Drug: Inter-Therapy - MEL-20+CFZ-TD-PACE (75%) — Melphalan (MEL) and Carfilzomib (CFZ) will be given into a central venous catheter. Thalidomide (T) is a capsule and Dexamethasone (D) is a pill; both will be taken by mouth. Cisplatin (P), Adriamycin (A), Cyclophosphamide (C) and Etoposide (E) are all given into the vein (IV) by a continuous infusion through a central catheter. After completion of the continuous chemotherapy, Granulocyte colony-stimulating factor (G-CSF), a shot just under the skin to help the bone marrow and blood counts recover more quickly after chemotherapy, will be given.
  Regimen: CFZ 27 mg/m2 on days 1-2; MEL 5 mg/m2/d, T 200 mg/d, D 20 mg/d, P 7.5 mg/m2/d, A 7.5 mg/m2/d, C 75 mg/m2/d, and E 60 mg/m2/d on days 1-4.
  Optional Bridging with T 50 mg/d and D 20 mg on day 1-4 every 21 days until 2nd transplant.
  Other Names: Melphalan (Alkeran™); Carfilzomib (Kyprolis®); Thalidomide (Thalomid®); Dexamethasone (Decadron®); Cisplatin (CDDP) (Platinol®); Doxorubicin (Adriamycin®); Cyclophosphamide (Cytoxan®); Etoposide (VP-16) (Vepesid®)
Drug: Second Transplant - MEL-80+CFZ-TD-PACE + PBSC (biologic) — Melphalan (MEL) and Carfilzomib (CFZ) will be given into a central venous catheter. Thalidomide (T) is a capsule and Dexamethasone (D) is a pill; both will be taken by mouth. Cisplatin (P), Adriamycin (A), Cyclophosphamide (C) and Etoposide (E) are all given into the vein (IV) by a continuous infusion through a central catheter. After completion of the continuous chemotherapy, Granulocyte colony-stimulating factor (G-CSF), a shot just under the skin to help the bone marrow and blood counts recover more quickly after chemotherapy, will be given.
  Regimen: CFZ 20 mg/m2 on days -5 & -4; MEL 20 mg/m2/d, T 200 mg/d, D 40 mg/d, P 10 mg/m2/d, A 10 mg/m2/d, C 100 mg/m2/d, and E 80 mg/m2/d on days -5 & -2; PBSC transplant on day 0.
  Optional Bridging with T 50mg/d and D 20 mg on day 1-4 every 21 days until consolidation.
  Other Names: Autologous Peripheral Blood Stem Cell Transplant; Melphalan (Alkeran™); Carfilzomib (Kyprolis®); Thalidomide (Thalomid®); Dexamethasone (Decadron®); Cisplatin (CDDP) (Platinol®); Doxorubicin (Adriamycin®); Cyclophosphamide (Cytoxan®); Etoposide (VP-16) (Vepesid®)
Drug: Consolidation - CFZ-TD-PACE — Carfilzomib (CFZ) will be given into a central venous catheter. Thalidomide (T) is a capsule and dexamethasone (D) is a pill; both will be taken by mouth. Cisplatin (P), adriamycin (A), cyclophosphamide (C) and etoposide (E) are all given into the vein (IV) by a continuous infusion through a central catheter.
  Regimen: CFZ 27 mg/m2 on days 1-2; T 200 mg/d, D 40 mg/d, P 7.5 mg/m2/d, A 7.5 mg/m2/d, C 300 mg/m2/d, and E 30 mg/m2/d on days 1-4.
  Other Names: Carfilzomib (Kyprolis®); Thalidomide (Thalomid®); Dexamethasone (Decadron®); Cisplatin (CDDP) (Platinol®); Doxorubicin (Adriamycin®); Cyclophosphamide (Cytoxan®); Etoposide (VP-16) (Vepesid®)
Drug: Maintenance - CFZ-R(T)-D — Carfilzomib (CFZ) will be given into a central venous catheter. Thalidomide (T) and lenalidomide (R) are capsules and dexamethasone (D) is a pill; all will be taken by mouth.
  Regimen: For Cycles 1-12 CFZ 27 mg/m2/wk and D 12 mg/wk on days 1, 8, 15, & 22; lenalidomide (R) 15 mg/d on days 1-21. For Cycles 13-24 CFZ 27 mg/m2/wk and D 12 mg/wk on days 1, 8, 15, & 22. T may be substituted for R at 100 mg/day at the treating physician's discretion.
  Other Names: Carfilzomib (Kyprolis®); Lenalidomide (CC-5013) (Revlimid®); Dexamethasone (Decadron®); Thalidomide (Thalomid®)

SUMMARY:
The purpose of this study is to improve the clinical outcomes of research subjects with high-risk multiple myeloma in the context of the immediately preceding Total therapy 5 trial 2008-02 and Total therapy 3 trials 2003-33 and 2006-66.

DETAILED DESCRIPTION:
Total therapy 5B will attempt to accelerate and sustain, at 2 years from starting therapy, the proportion of subjects in complete remission by reducing host-imposed toxicity and facilitating timely completion of highly synergistic 8-drug combination therapy, including the next generation proteasome inhibitor, Carfilzomib. This will result in avoiding multiple myeloma re-growth that, we postulate, ensued in Total therapy 3 during recovery phases from severe de-conditioning. It is speculated that the incidence of positive minimal residual disease will be reduced with the addition of one cycle of consolidation therapy. The following approach will be implemented:

* apply a 4-day fractionated lower dose melphalan (80 mg/m2) together with CFZ-TD-PACE regimen in MEL80-CFZ-TD (carfilzomib, thalidomide, dexamethasone) PACE as a hopefully less toxic and more effective transplant regimen
* interspersed with 1 cycle of non-transplant supported MEL-20-CFZ-TD (carfilzomib, thalidomide, dexamethasone) PACE (in lower doses than with transplant) inter-therapy (reduced from two cycles due to prolonged thrombocytopenia)
* followed by CFZ-TD (carfilzomib, thalidomide, dexamethasone) PACE consolidation therapy post transplant #2
* CFZ-RD (carfilzomib, lenalidomide and dexamethasone) maintenance for 1 year followed by CFZ-D for an additional year

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed active MM requiring treatment. Patients with a previous history of smoldering myeloma will be eligible if there is evidence of progressive disease requiring chemotherapy.
* Patients must be either untreated or have not had more than one cycle of systemic MM therapy, excluding bisphosphonates and localized radiation.
* Participants must have high-risk disease, as defined by GEP70 risk score of ≥ 0.66
* Zubrod ≤ 2, unless solely due to symptoms of MM-related bone disease.
* Patients must have a platelet count of ≥ 50,000/μL, unless lower levels are explained by extensive bone marrow plasmacytosis.
* Patients must be at least 18 years of age and not older than 75 years of age at the time of registration.
* Participants must have preserved renal function as defined by a serum creatinine level of < 3 mg/dL.
* Participants must have an ejection fraction by ECHO or MUGA scan ≥ 45%
* Patients must have adequate pulmonary function studies > 50% of predicted on mechanical aspects (FEV1, FVC, etc) and diffusion capacity (DLCO) > 50% of predicted. If the patient is unable to complete pulmonary function tests due to MM related pain or condition, exception may be granted if the principal investigator documents that the patient is a candidate for high dose therapy.
* Patients must have signed an IRB-approved informed consent indicating their understanding of the proposed treatment and understanding that the protocol has been approved by the IRB.

Exclusion Criteria:

* Does not have high-risk disease
* Poorly controlled hypertension, diabetes mellitus, or other serious medical illness or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Patients must not have prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has not received treatment for one year prior to enrollment. Other cancers will only be acceptable if the patient's life expectancy exceeds five years.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Subjects of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06-10 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frits Van Rhee, MD, Ph.D, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pawlyn C. High-risk myeloma: a challenge to define and to determine the optimal treatment. Lancet Haematol. 2021 Jan;8(1):e4-e6. doi: 10.1016/S2352-3026(20)30361-6. Epub 2020 Dec 22. No abstract available. PMID 33357481
- [Derived] Davies FE, Rosenthal A, Rasche L, Petty NM, McDonald JE, Ntambi JA, Steward DM, Panozzo SB, van Rhee F, Zangari M, Schinke CD, Thanendrarajan S, Walker B, Weinhold N, Barlogie B, Hoering A, Morgan GJ. Treatment to suppression of focal lesions on positron emission tomography-computed tomography is a therapeutic goal in newly diagnosed multiple myeloma. Haematologica. 2018 Jun;103(6):1047-1053. doi: 10.3324/haematol.2017.177139. Epub 2018 Mar 22. PMID 29567784

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Treatment: MEL-CFZ-TD-PACE: Melphalan and Carfilzomib will be given into a central venous catheter. Dexamethasone is a pill that is taken by mouth daily for 4 days. Thalidomide is a capsule taken by mouth for 4 days. Cisplatin, Adriamycin, Cyclophosphamide and Etoposide are all given into the vein (IV) by a continuous infusion through a central catheter for 4 days. After completion of the four days of continuous chemotherapy, a drug G-CSF will be given. This is a shot just under the skin to help the bone marrow and blood counts recover more quickly after chemotherapy.
Period: Overall Study
Arm/Group | Study Treatment
Started | 20
Completed | 1
Not Completed | 19

BASELINE CHARACTERISTICS:
Arm/Group | Study Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63.5 [44.4 to 69.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: The Remission Rate for Participants With High-risk Myeloma
Description: Toward improving the clinical outcomes of research subjects with high-risk MM (HR-MM) in the context of the immediately preceding TT5 trial 2008-02 and TT3 trials 2003-33 and 2006-66, TT5B will attempt to accelerate and sustain, at 2 years from starting therapy, the proportion of subjects in complete remission (AS-CR-2) by reducing host-imposed toxicity and thus facilitating timely completion of highly synergistic 8-drug combination therapy, including the next generation proteasome inhibitor, Carfilzomib (CFZ). This will result in avoiding MM re-growth that, we postulate, ensued in TT3 during recovery phases from severe de-conditioning. Furthermore, we speculate that the incidence of positive minimal residual disease (MRD) will be reduced with the addition of one cycle of consolidation therapy.
Time Frame: from baseline to either death or study completion for each subject (up to approximately 48 months)
Population: Nineteen (19) subjects discontinued study prior to completion. Only one (1) subject completed all study related activities.
Measure: Number; unit: Participants
Groups:
- Total Therapy 5B: Induction 1 - MEL-10+CFZ-TD-PACE, Optional Bridging with TD, First Transplant - MEL-80+CFZ-TD-PACE + PBSC, Optional Bridging with TD, Inter-Therapy - MEL-20+CFZ-TD-PACE (75%), Optional Bridging with TD, Second Transplant - MEL-80+CFZ-TD-PACE + PBSC, Optional Bridging with TD, Consolidation - CFZ-TD-PACE, Maintenance - CFZ-R(T)-D
Arm/Group | Total Therapy 5B
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Time Frame: From baseline to either death or study completion for each subject (up to 48 months)
Arm/Group | Study Treatment
All-Cause Mortality (participants affected / at risk) | 4/20
Serious Adverse Events (participants affected / at risk) | 13/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Treatment (N=20)
Hospitalization for Syncope (Cardiac disorders) | 1 (1)
Hospitalization for Parainfluenza (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization for Hematuria (Blood and lymphatic system disorders) | 1 (1)
Hospitalization for K. Pneumonia UTI (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization for Neutropenic Colitis (Gastrointestinal disorders) | 1 (1)
Colitis / Grade 3 (Gastrointestinal disorders) | 1 (1)
Leukopenia / Grade 2 (Immune system disorders) | 1 (1)
Neutropenia / Grade 3 (Immune system disorders) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hospitalization for Uncontrolled Pain (General disorders) | 1 (1)
Hospitalization for Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization for Sinus Bradycardia (Cardiac disorders) | 1 (1)
Hospitalization for Atrial Fibrillation (Cardiac disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization for Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Hospitalization for Chest Pain (General disorders) | 1 (1)
Hospitalization Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalization for L. hip pain (Injury, poisoning and procedural complications) | 1 (1)
Myelodysplastic Snydrome (MDS) (Blood and lymphatic system disorders) | 1 (1)
Acute Myeloid Leukemia (AML) (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Study Treatment (N=20)
Anemia (Blood and lymphatic system disorders) | 20
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 9
Lymphocyte count decreased (Blood and lymphatic system disorders) | 20
Neutrophil count decreased (Blood and lymphatic system disorders) | 19
Platelet count decreased (Blood and lymphatic system disorders) | 20
Wbc decrease (leukopenia) (Blood and lymphatic system disorders) | 20
Atrial fibrillation (Cardiac disorders) | 2
Cardiac disorders - other (Cardiac disorders) | 4
Heart failure (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 8
Sinus tachycardia (Cardiac disorders) | 8
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Vestibular Disorder (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 2
Dry eye (Eye disorders) | 1
Eye disorders - Other, (Eye disorders) | 1
Floaters (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 5
Anal hemorrhage (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 4
Colitis (Gastrointestinal disorders) | 2
Colonic perforation (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 18
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 6
Enterocolitis (Gastrointestinal disorders) | 1
Esophageal obstruction (Gastrointestinal disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5
Gastrointestinal disorders - Other, (Gastrointestinal disorders) | 4
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastroparesis (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 20
Oral pain (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 4
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 8
Edema face (General disorders) | 5
Edema limbs (General disorders) | 14
Edema trunk (General disorders) | 2
Fatigue (General disorders) | 18
Fever (General disorders) | 10
Flu like symptoms (General disorders) | 2
Gait disturbance (General disorders) | 4
Malaise (General disorders) | 1
Neck edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 6
Pain (General disorders) | 11
Alanine aminotransferase increased (Hepatobiliary disorders) | 15
Alkaline phosphatase increased (Hepatobiliary disorders) | 16
Aspartate aminotransferase increased (Hepatobiliary disorders) | 14
Blood bilrubin increased (Hepatobiliary disorders) | 7
Hypoalbuminemia (Hepatobiliary disorders) | 20
Allergic reaction (Immune system disorders) | 1
Immune system disorders - Other, (Immune system disorders) | 6
Abdominal infection (Infections and infestations) | 1
Infections and infestations - Other, (Infections and infestations) | 11
Lung infection (Infections and infestations) | 5
Otitis media (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Rhinitis infective (Infections and infestations) | 7
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Ejection fraction decreased (Investigations) | 1
Weight gain (Investigations) | 9
Anorexia (Metabolism and nutrition disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 20
Hyperkalemia (Metabolism and nutrition disorders) | 7
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 20
Hypokalemia (Metabolism and nutrition disorders) | 16
Hypomagnesemia (Metabolism and nutrition disorders) | 20
Hyponatremia (Metabolism and nutrition disorders) | 20
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 10
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Ataxia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 11
Dysgeusia (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 9
Myelitis (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 14
Presyncope (Nervous system disorders) | 2
Sinus pain (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 8
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 11
Acute kidney injury (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Creatinine increased (Renal and urinary disorders) | 15
Hematuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 6
Urinary retention (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 12
Apnea (Respiratory, thoracic and mediastinal disorders) | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 6
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 3
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6
Dermatology/skin - bruising (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Skin and subcutaneous tissue disorders - Other, (Skin and subcutaneous tissue disorders) | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Social circumstances - Other, (Social circumstances) | 5
Flushing (Vascular disorders) | 3
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 13
Hypotension (Vascular disorders) | 14
Thromboembolic event (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to futility as determined by Amgen's Carfilzomib NASCR program in addition to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT02128230/Prot_SAP_000.pdf